CLINICAL TRIAL: NCT07220122
Title: Impact of Exogenous Ketones on Sleep and Breathing in Healthy Volunteers
Brief Title: Impact of Exogenous Ketones on Breathing in Healthy Volunteers
Acronym: K-BREATHE
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00517978-2
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
Keywords: ketones breathing exogenous
MeSH Terms: interventions — 1,3-butylene glycol

STUDY DESIGN:
Intervention Model Description: Single blind placebo controlled randomized crossover design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketones first (Experimental): Visit 1: ketones, Visit 2: Placebo
  Interventions: Dietary Supplement: 1,3 butanediol; Dietary Supplement: Placebo
- Placebo first (Experimental): Visit 1: Placebo, Visit 2: ketones
  Interventions: Dietary Supplement: 1,3 butanediol; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 1,3 butanediol — 40 mg Ketone-IQ beverage
Dietary Supplement: Placebo — Placebo (taste matched)

SUMMARY:
Exogenous ketones (EK) are compounds that can increase the level of ketones in the body without needing to change what an individual eats.

Although EK have been researched mainly in relation to energy and exercise, there haven't been many studies focusing specifically on how EKs affect breathing using well-established scientific methods. The investigators believe that EK may help improve breathing, which could be beneficial for situations like high altitudes, sleep apnea, and exercise.

To explore how EK might influence breathing, the investigators are conducting a randomized, placebo-controlled crossover study with healthy volunteers.

DETAILED DESCRIPTION:
Healthy volunteers will undergo daytime hypercapnic ventilatory response (HCVR) testing before and after ingesting 40g of exogenous ketones or placebo. Circulating ketone levels (beta-hydroxybutyrate) will be measured at baseline, 1 hour, and 2.5 hours after ingestion (immediately before HCVR testing). Studies will require two visits with a minimum of 48 hr. (and up to a max of 14 days) of washout.

The specific ketone product to be tested is 1,3 butanediol (1,3BD) in a commercially available formulation called "Ketone IQ". A taste-matched placebo will also be supplied by the sponsor. 1,3BD is converted by liver metabolism into the ketone body beta-hydroxybutyrate (BHB) and has been utilized in multiple studies.

PROCEDURES:

This is a randomized, single-blind, crossover study. Each participant will complete two testing sessions with a minimum of 48-hour washout period between visits. The single-blind design enables research staff to measure BHB levels and assess pharmacokinetic timing for potential adjustments to procedure timing, while keeping participants blinded to the intervention.

Baseline visit: A medical history and physical examination will be performed. A urine pregnancy screening test will be conducted for women under 60 years of age. A "run-in" procedure will be performed to confirm that participants can tolerate the taste of the ketone supplement. Participants will then be randomized to one of two arms:

* Group A: Visit 1 Ketones, Visit 2 Placebo
* Group B: Visit 1 Placebo, Visit 2 Ketones

Session 1:

HCVR Procedure: Participants will wear a facemask connected to a breathing circuit with a three-way stopcock, allowing inhaled gas to be switched from ambient air to a pre-mixed gas source. A one-way valve will divert exhaled gas to prevent rebreathing. The participant will breathe room air for 3-5 minutes to collect baseline ventilation data. The investigators will then switch to a non-diffusing gas bag containing 7% Carbon Dioxide (CO₂) / 93% O₂ and the participant will breathing this hypercapnic gas until end-tidal CO₂ (ETCO₂) reaches a stable plateau and is maintained (up to 3 minutes, as tolerated).

Exhaled CO₂ and airflow will be continuously monitored using a pneumotachograph to derive tidal volume and respiratory rate. The HCVR slope will be calculated as minute ventilation (L/min) plotted against end-tidal CO₂ (mmHg).

Session Sequence:

1. Participants will arrive at the lab after an overnight fast.
2. Baseline HCVR testing will be conducted before study product ingestion.
3. Participants will ingest 40 g Ketone-IQ or placebo.
4. Repeat HCVR testing 2.5 hours post-ingestion.

Capillary BHB levels will be measured at baseline, 1 hour, and 2.5 hours post-ingestion of Ketone-IQ. Participants will not see the BHB levels (so that the placebo condition will be appropriately masked).

Session 2:

This session will mirror Session 1, with participants crossing over to the alternate condition (i.e., Ketone-IQ or placebo), following a minimum 48-hour washout period.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18 - 30 kg/m2

Exclusion Criteria:

* No concomitant sleep disorder (e.g. sleep apnea, insomnia, restless leg syndrome, narcolepsy, idiopathic hypersomnia). If there is no known diagnosis of sleep apnea, a STOP-BANG score of 5 or higher is an exclusion.
* No current daytime respiratory impairment such as uncontrolled asthma, or uncontrolled Chronic Obstructive Pulmonary Disease (COPD), pneumonia, interstitial lung disease.
* No known history of chronic renal disease or diabetes (type 1 or type 2).
* No use of supplemental oxygen.
* Cannot be on a low carbohydrate (<130 g carbohydrate/day) or ketogenic diet, intermittent fasting, or consuming exogenous ketones
* Cannot be pregnancy or breastfeeding
* Cannot be on medications: acetazolamide or Sodium-glucose cotransporter-2 (SGLT2) inhibitor, daily opioid use.
* No history of claustrophobia or panic disorder
* No frequent alcohol intake (more than 1 drink per day on average, or > 10 drinks per week).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Hypercapnic Ventilatory Response (HCVR) | During each visit, one measurement at baseline, repeated again 2.5 hours after ingesting Ketone-IQ or Placebo
  Minute ventilation (L/min) while breathing 7% Carbon Dioxide (CO2). Measured once during each visit.

SECONDARY OUTCOMES:
Ketone Level | During each visit measured 4 times (baseline, 1 hour, 2.5 hours post-ingestion)
  Beta-hydroxybutyrate (BHB) in millimole (mmol) from blood. Measured 4 times during each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request de-identified primary data related to ketone levels and breathing responses will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: 3 years following study completion.
Access Criteria: Researchers requesting access must contact the PI for permission.